CLINICAL TRIAL: NCT02191839
Title: Single Dose Administration of Alpha-1 Anti-Trypsin for the Amelioration of Organ Injury and Post Operative Bleeding in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass: Double-blind, Placebo-controlled Pilot Study
Brief Title: Single Dose Administration of Alpha-1 Anti-Trypsin for the Amelioration of Organ Injury in Patients Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Dan Abramov, Dr, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOR 133-13 ctil
Record Dates: First submitted 2014-07-07; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Post Cardiac Surgery Systemic Inflammatory Response
Keywords: cardiac surgery; alpha 1 antitrypsin; inflammation; post operative bleeding; organ function
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Inflammation | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha 1 antitrypsin (Active Comparator): patients receive 4 grams of IV alpha 1 antitrypsin preoperatively
  Interventions: Drug: Alpha 1-Antitrypsin
- placebo (Placebo Comparator): 10 patients will randomely receive placebo

INTERVENTIONS:
Drug: Alpha 1-Antitrypsin
  Arms: alpha 1 antitrypsin

SUMMARY:
Protocol Summary STUDY DESIGN A pilot, prospective, double blind, randomized, placebo controlled study.

STUDY POPULATION Patients assigned to elective CABG with cardiopulmonary bypass (CPB) at the Department of Cardiothoracic Surgery, Soroka University Medical Center.

OBJECTIVE To evaluate anti-inflammatory effects, effects on organ function preservation, and postoperative blood loss reduction following AAT-1 administration in patients undergoing CABG with CPB.

PRIMARY ENDPOINT Postoperative organ function preservation and blood loss following preoperative single-dose AAT-1 administration.

SAMPLE SIZE CONSIDERATIONS A cohort of 20 patients will be recruited. Patients will be randomized to receive either AAT-1 or placebo prior to surgery. Whereas this is a proof of concept pilot study, statistical significance is not the primary objective.

INCLUSION CRITERIA 1. The study population will comprise patients between 40 and 70 years of age, irrespective of gender, at low or intermediate operative risk (calculated Logistic Euroscore stratification of 5% or less), assigned to elective CABG with CPB. Recruitment depending on patients informed consent.

EXCLUSION CRITERIA Co-existing conditions including:

1. Coagulation abnormalities
2. Severe pulmonary disease defined by blood oxygen saturation of 90% or less or FEV1 of less than 60% of predicted.
3. Renal dysfunction defined be serum creatinine levels higher or equal to 1.8 mg%,
4. Abnormal liver function tests
5. Uncontrolled diabetes mellitus,
6. Severe peripheral vascular disease
7. Prior cerebrovascular neurological event.
8. Abnormal left or right ventricular function.
9. Treatment with warfarin or thienopyridine class of anti platelet agents.

DETAILED DESCRIPTION:
3 Background The use of cardiopulmonary bypass (CPB) during cardiac surgery elicits generalized non-specific systemic inflammatory response syndrome (SIRS) and subsequent activation of the cytokine, complement, and coagulation-fibrinolytic cascades (1). In approximately 11% of the patients SIRS may deteriorate to severe multi-organ failure (MOF) resulting in mortality rate of 40-98%.

Inflammatory modulation by intraoperative administration of anti-inflammatory substances has been advocated to attenuate the effects of SIRS. Attempts have subsequently focused on aprotinin which inhibits proteases that are key mediators in the complement, coagulation, and fibrinolytic system. Related anti-inflammatory properties of aprotinin include the inhibition of platelets, neutrophils and kallikrein activation. Reduction in blood loss and reduced need for allogenic blood transfusions have been proposed as additional mechanisms by which aprotinin limits the inflammatory response (2). The use of aprotinin during cardiac surgery, however, was discontinued following alarming results in terms of higher rate of bypass graft occlusion and overall inferior postoperative outcome.

AAT-1 mechanism of action:

Similar to aprotinin, α1-Antitrypsin (AAT) is a 52-kDa circulating serine protease inhibitor classified as a SERPIN protein. Besides its ability to inhibit serine proteases, accumulating data suggest that AAT-1 possesses independent anti-inflammatory and tissue-protective effects (3). AAT-1 modifies dendritic cell maturation and promotes regulatory T-cell differentiation, induces interleukin (IL)-1 receptor antagonist and IL-10 release, protects various cell types from cell death, inhibits caspases-1 and -3 activities and inhibits IL-1 production and activity (4). Contradictory to classic immunosuppressants, AAT-1 allows undeterred isolated T-lymphocyte responses (5).These effects have been repeatedly corroborated.

Unlike aprotinin, AAT-1 is produced from human plasma, and does not have strong pro coagulant characteristics.

AAT-1 in different clinical settings:

Circulating AAT-1 levels increase by 4-fold during acute-phase response (3). Patients with low circulating levels of AAT-1 are at increase risk for lung, liver and pancreatic destructive diseases, particularly emphysema (3). Preclinical and clinical studies have shown that AAT-1 therapy for non-deficient individuals is safe, and may modify disease progression in type 1 and type 2 diabetes, acute myocardial infarction, rheumatoid arthritis, inflammatory bowel disease, cystic fibrosis, transplant rejection, graft versus host disease and multiple sclerosis (6-17, 32,33,37,38) . AAT-1 treatment has subsequently advanced from replacement therapy to potential treatment for a broad spectrum of inflammatory and immune-mediated diseases. AAT-1 also appears to be antibacterial and an inhibitor of viral infections, such as influenza and human immunodeficiency virus (HIV) (18).

Human pharmacokinetic data:

In patients with AAT-1 deficiency, intravenous administration of AAT-1 in a dose of 60 mg per kg body weight maintain plasma levels resembling acute phase response immediately after administration, and retain an appropriate level of serum AAT above the protective threshold (50 mg/dl) a week afterwards (39).

Rational of AAT-1 dosage:

Based on previous studies and clinical practice, the administration of multiple intravenous dosage of 60 mg per kg body weight of AAT-1 is safe and is associated with low incidence of benign side-effects.

Derived from pharmacokinetic studies (39), AAT-1 plasma levels immediately following the administration of this external dosage resembles acute phase response. A 30% reduction in AAT-1 plasma levels is anticipated with gradual return to preoperative levels after termination of CPB (40).

Risk/ benefit of the study:

The role of AAT-1 in mitigating inflammatory response has been established. CPB is a potent stimulator of inflammatory cascades and associated with bleeding diatheses, coagulation abnormalities, potentially leading to organ dysfunction. To date, the administration of AAT-1 in patients undergoing cardiac surgery with CPB has not been explored. It may be postulated that inherent AAT-1 effects may offset deleterious CPB effects. This may clinically result in improved preservation of organ function, reduced postoperative bleeding and reduced hospital stay. The benefits of other protease inhibitors in corresponding settings have been recently demonstrated (41-43).

As mentioned above, administration of AAT-1 in various clinical settings is considered safe with low rate of side effects (see section 6.1 - potential risks).

4 Methods 4.1 Primary Objective

1. To evaluate the efficacy and safety of preoperative AAT-1 administration in patients undergoing CABG with CPB.
2. Postoperative blood loss and organ function will be assessed.

To date, no data exists with regard to AAT-1 effects in the settings of CPB. The primary goals of this study are to evaluate anti-inflammatory effects, organ function preservation (1-2) and postoperative blood loss reduction following AAT-1 administration in patients undergoing cardiac surgery with CPB.

4.2 Determination of Study Eligibility 4.2.1 Inclusion Criteria

1. Male/female patients 40-70 years of age.
2. Candidates for isolated CABG with CPB.
3. Calculated logistic Euroscore risk stratification of 5% or less.
4. Signed patient's written informed consent.

4.2.2 Exclusion Criteria

Co-existing conditions including:

10. Coagulation abnormalities 11. Severe pulmonary disease defined by blood oxygen saturation of 90% or less or FEV1 of less than 60% of predicted.

12. Renal dysfunction defined be serum creatinine levels higher or equal to 1.8 mg%, 13. Abnormal liver function tests 14. Uncontrolled diabetes mellitus, 15. Severe peripheral vascular disease 16. Prior cerebrovascular neurological event. 17. Abnormal left or right ventricular function. 18. Treatment with warfarin or thienopyridine class of anti-platelet agents. 4.2.3 Withdrawal Criteria Patients will preserve the right to withdraw from the study at any time during treatment without prejudice.

If medically indicated, the principal investigator or the surgeon poses the right to discontinue patient enrollment at any stage of the study.

Discontinuation (failure to complete the study) will be documented. The reason for discontinuation will be recorded.

Potential causes that may lead to discontinuation include:

* Adverse event(s)
* Protocol violation
* Patient withdrew consent
* Administrative problems 4.3 Enrollment Prior to participation in this study, the Investigator will obtain written appropriate approval for the protocol and the informed consent form the Ethics Committee (EC) and other local regulatory organizations. The approved consent form will clearly reflect the EC approval date.

Failure to obtain a signed and hand dated informed consent prior to the procedure constitutes a protocol violation, and subsequently reportable to the EC.

4.4 Subject Screening Patients that have been already scheduled for isolated CABG operation will be addressed by a member of the research team during the preoperative waiting period (either in the Department of Cardiothoracic Surgery, the Department of Cardiology or the Department of Internal Medicine). The goal of the study, procedure and incentive will be explained by a research staff member to each potential participant. Consenting subjects will be asked to provide written consent.

4.4.1 Randomization The study participants will be randomized to receive either single dose AAT-1 60 mg per kg or placebo.

4.4.2 Trial medication administration: Preparation and dosing of AAT-1 will be performed by an unblinded pharmacist. The medication will be diluted just prior to administration. The placebo solution will comprise human albumin that resembles the color and consistency of AAT-1 solution. The medication will be given 3-5 hours prior to surgery (skin incision). Administration rate of the drug will not exceed 0.04 ml per kg per minute (approximately 60-80 minutes). Vital signs including blood pressure, pulse rate and body temperature will be correspondingly monitored.

The patients, research staff, laboratory personnel and data analysts will remain blinded to the identity of the treatment from the time of randomization and until database lock. Data unblinding will commence in the case of patient's emergency.

A randomization list will be produced by the pharmacist, however, will be secured and confidential until time of unblinding.

4.4.3 Surgical technique Consistent with our routine policy, fentanyl citrate (20-50mcg/kg), midazolam (2-3mg) and isoflurane (0.5-2%) will be used for induction and maintenance of anesthesia.

Standard median sternotomy will be followed by procurement of the conduits. Heparin loading dose will be administered to achieve a kaolin activated coagulation time (ACT). Ascending aorta - right atrial cannulation will be performed to institute CPB and ACT will be monitored at 480 seconds or more. Standard centrifugal pump and a membrane oxygenator will be used for extracorporeal circulation (cardiopulmonary bypass). Compatible with the standard technique, systemic active cooling will be avoided and patients core temperature will remain range between 32 and 37˚C. Distal anastomoses will be performed during single aortic cross-clamp and blood cardioplegic arrest. Proximal anastomoses will be performed during aortic cross-clamp. Cold (10˚C) blood cardioplegic solution will be delivered in a 4:1 ratio. Cardioplegia will be delivered antegrade via the aortic root with or without additional retrograde administration via the coronary sinus. After cardioplegic induction (10 ml / Kg), intermittent doses (300 - 500 ml) will be administered following completion of each distal anastomosis. Heparin will be reversed using protamine sulphate in a ratio of 1:1 after weaning from CPB.

4.4.4 Data collection Preoperative data: Demographic, morphological and clinical descriptors including age, gender, body mass index (BMI), body surface area (BSA) co-morbidity, Euroscore risk-stratification, medication, etc. will be recorded. Preoperative laboratory analysis will include complete blood count, coagulation profile, serum creatinine levels and creatinine clearance, liver function test and arterial blood gases test and serology for HIV,HCV,HBC. Compatible with our routine policy, all patients will undergo preoperative echocardiography, coronary angiography, chest x-ray, lung function tests (spirometry) and carotid artery duplex study.

Study participants will be assigned to undergo preoperative brain MRI; subjected to the protocol described below.

Intraoperative: The type of surgery will be classified. The following data will be recorded: heparin dose given prior to bypass initiation; activated clotting time (ACT) counts during the operation (prior, during and after CPB); operative time, cross-clamp time and CPB time; number of trials to wean from CPB, type of inotropes and dosage used during weaning from CPB; blood products utilization during surgery. Allergic reactions or adverse events observed by the surgeon or anesthesiologist will be documented. The individual surgeon's impression regarding bleeding tendency will be recorded.

Postoperative organ function and blood loss evaluation:

The occurrence and magnitude of systemic inflammatory response and organ dysfunction will be recorded and quantified by laboratory markers. Related laboratory markers will be monitored on a daily basis during the recovery period (in the intensive care unit and at the ward). The following organs and corresponding markers will be monitored:

Pulmonary function: Pulmonary function will be evaluated by measured overall mechanical ventilation time, peak inspiratory pressures (PIP), plateau pressures, physiologic dead space and static and dynamic lung compliance. Bronchoalveolar lavage (BAL) will be performed 3 hours after operation (while the patient is anesthesized and intubated) and extracted fluid will be analyzed for inflammatory markers. A-a DO2 calculation [AaDO2 = (713 x FiO2) - (pCO2 / 0.8) - (paO2)] will be measured daily.

Complete pulmonary function test will be performed before and 4 days after the operation. Chest radiographs will be evaluated and quantified by an independent radiologist for the occurrence of atelectasis, pulmonary edema, or pleural changes.

Renal function: Daily measurements of urine output, serum creatinine levels, creatinine clearance and urinary albumin levels. Acute kidney injury (AKI) markers will be sampled in the ICU.

Brain injury assessment: The degree of insult to the brain will be measured by plasma S-100 proteinlevels. Assessment of damage to the blood-brain barrier (BBB) will be performed by magnetical resonance imaging (MRI) modality (see technique protocol below).

Hepatic function: Daily measurements of serum hepatic enzymes levels. Cardiac function: Monitoring of cardiac enzymes levels; need and magnitude of required inotrope treatment; occurrence of low cardiac output syndrome (defined as systolic blood pressure of 90 mmHg or less coupled with central venous pressure (CVP) of 15 mmHg or more) and incidence of cardiac arrhythmias. Transthoracic echocardiography examination will be performed on postoperative day 5 and assessed by an independent cardiologist.

Blood loss: Operative and postoperative blood loss will be monitored as well as daily hemoglobin levels. Daily platelet counts and thromboelastograms will be performed. The distribution of blood products and total administered will be recorded daily. Postoperative CRP levels will be evaluated daily.

Blood sampling and laboratory analysis methods for cytokine levels:

Ten mL whole blood venous EDTA samples will be collected from radial artery catheter at five specified occasions: before induction of anaesthesia, 30 minutes after aortic cross-clamp positioning and 3, 6, and 9 hours after aortic cross clamp positioning. The blood samples will be subsequently centrifuged at 4 °C for 15 min and the serum stored at -70 °C. Samples will be analyzed for the following markers: Polimorphonuclear Neutrophil Elastase (PMNE), Interleukin-1α (IL-1α), Interleukin-1ß (IL-1ß), Interleukin-2 (IL-2), Interleukin-4 (IL-4), Interleukin-6 (IL-6), Interleukin-8 (IL-8), Interleukin-10 (IL-10), Interferon-γ (IFN-γ), Tumor Necrosis Factor-α (TNF-α), Vascular Endothelial Growth Factor (VEGF), Monocyte Chemoattractant Protein-1 (MCP-1), and Endothelial Growth Factor (EGF).

Daily blood samples will be collected postoperatively for platelet count, renal function, liver function, CRP levels S-100 protein and troponin.

Early postoperative adverse events will be documented. These include 30-day mortality, new neurological events, myocardial infarction, renal dysfunction, need for re-exploration for bleeding and deep sternal wound infection.

Blood-Brain Barrier (BBB) assessment by MRI The imaging modality used for BBB assessment will be MRI scanner (Philips 3T or General Electric 1.5T). The examination format will include 24 cm FOV, 35 contiguous interleaved slices, 3.5-4 mm thick and co-localized across series. Trace-weighted DWI images will be obtained at b=1000 from a 13-15 direction DTI sequence with an in-plane resolution of 2.5×2.5mm and TR/TE=10s/58ms at 3T or TR/TE=10s/72ms at 1.5T. T2-FLAIR images will be obtained with an in-plane resolution of 0.94×0.94 mm, TR/TE=9000/120 ms and TI=2600 ms at 3T or TR/TE=9000/140 ms and TI=2200 ms at 1.5T. (25)

ELIGIBILITY:
Inclusion Criteria:

1. The study population will comprise patients between 40 and 70 years of age, irrespective of gender, at low or intermediate operative risk (calculated Logistic Euroscore stratification of 5% or less), assigned to elective CABG with CPB. Recruitment depending on patients informed consent.

Exclusion Criteria:

Co-existing conditions including:

1. Coagulation abnormalities
2. Severe pulmonary disease defined by blood oxygen saturation of 90% or less or FEV1 of less than 60% of predicted.
3. Renal dysfunction defined be serum creatinine levels higher or equal to 1.8 mg%,
4. Abnormal liver function tests
5. Uncontrolled diabetes mellitus,
6. Severe peripheral vascular disease
7. Prior cerebrovascular neurological event.
8. Abnormal left or right ventricular function.
9. Treatment with warfarin or thienopyridine class of anti platelet agents -

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
post operative inflammatory response | post operative day 1-5
  1. The occurrence and magnitude of systemic inflammatory response and organ dysfunction will be recorded and quantified by laboratory markers. Related laboratory markers will be monitored on a daily basis during the recovery period (in the intensive care unit and at the ward).
Pulmonary function: | post op day 1-5
  Pulmonary function will be evaluated by measured overall mechanical ventilation time, peak inspiratory pressures (PIP), plateau pressures, physiologic dead space and static and dynamic lung compliance. Bronchoalveolar lavage (BAL) will be performed 3 hours after operation (while the patient is anesthetised and intubated) and extracted fluid will be analyzed for inflammatory markers. A-a DO2 calculation [AaDO2 = (713 x FiO2) - (pCO2 / 0.8) - (paO2)] will be measured daily.
  Complete pulmonary function test will be performed before and 4 days after the operation. Chest radiographs will be evaluated and quantified by an independent radiologist for the occurrence of atelectasis, pulmonary edema, or pleural changes.
Renal function: | post op day 1-5
  Daily measurements of urine output, serum creatinine levels, creatinine clearance and urinary albumin levels. Acute kidney injury (AKI) markers will be sampled in the ICU.
Brain injury assessment: | post op day 1-5
  The degree of insult to the brain will be measured by plasma S-100 proteinlevels. Assessment of damage to the blood-brain barrier (BBB) will be performed by magnetical resonance imaging (MRI) modality
Hepatic function: | post op day 1-5
  Daily measurements of serum hepatic enzymes levels.
Cardiac function: | post op day 1-5
  Monitoring of cardiac enzymes levels; need and magnitude of required inotrope treatment; occurrence of low cardiac output syndrome (defined as systolic blood pressure of 90 mmHg or less coupled with central venous pressure (CVP) of 15 mmHg or more) and incidence of cardiac arrhythmias. Transthoracic echocardiography examination will be performed on postoperative day 5 and assessed by an independent cardiologist.
Blood loss: | post op day 1-2
  Operative and postoperative blood loss will be monitored as well as daily hemoglobin levels. Daily platelet counts and thromboelastograms will be performed. The distribution of blood products and total administered will be recorded daily. Postoperative CRP levels will be evaluated daily.

CONTACTS AND LOCATIONS:
Overall Officials: DAN ABRAHAMOV, DR, Principal Investigator — Soroka University Medical Center